CLINICAL TRIAL: NCT01693978
Title: Incentivizing Adherence to Prolonged Exposure With Substance Users
Brief Title: Contingency Outcomes in Prolonged Exposure
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jessica Peirce, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA032689-01A1 (NIH)
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Posttraumatic Stress Disorder; Substance Use Disorder
Keywords: PTSD; Prolonged Exposure; Comorbidity; Treatment; Methadone Maintenance; Substance Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reinforced Prolonged Exposure (RPE) (Experimental): All participants will be scheduled to attend a weekly Prolonged Exposure therapy session for 12 consecutive weeks, and followed for 12 additional weeks. RPE participants will receive voucher-based reinforcement contingent on attendance to scheduled Prolonged Exposure therapy sessions.
  Interventions: Behavioral: Prolonged Exposure Therapy; Behavioral: Voucher-Based Reinforcement
- Standard Prolonged Exposure (SPE) (Active Comparator): All participants will be scheduled to attend a weekly Prolonged Exposure therapy session for 12 consecutive weeks, and followed for 12 additional weeks.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Prolonged Exposure Therapy is considered the "gold standard" treatment for PTSD in psychiatry. It uses a cognitive-behavioral approach that repeatedly and systematically exposes patients to memories of their traumatic events to reduce fear and arousal. The PE therapy offered in this study will be based on procedures used by Foa and colleagues, described in their book-length treatment manual (Foa, Hembree, & Rothbaum, 2007).
  Other Names: PE Therapy
Behavioral: Voucher-Based Reinforcement — Those in the PE+CM condition will also be able to earn voucher-based incentives for each therapy session that they attend as scheduled, with a maximum of $480 for full adherence to all sessions. Specifically, participants will earn $30 for attending Session 1, $40 for attending Session 2, $50 for attending Session 3, and $60 for attending Sessions 4 through 9. There will be no payment for Sessions 10 through 12. Because it is very important that participants attend sessions on schedule, voucher values will be reset starting from $30 if participants miss a scheduled session. Vouchers can be exchanged for goods and services in the community (e.g., gift cards to local retailers).
  Other Names: Vouchers
  Arms: Reinforced Prolonged Exposure (RPE)

SUMMARY:
The aim of this research is to assess whether Contingency Management is effective in improving treatment adherence in substance use disordered (SUD) patients with comorbid PTSD. Although Prolonged Exposure therapy (PE) is the gold standard treatment for PTSD, the few studies of this treatment in substance users have shown poor adherence. Contingency Management is a well-established approach that could be used to enhance adherence to PE. From a consented sample of 125 opioid-dependent and methadone-treated patients at Addiction Treatment Services, an intent-to-treat sample of 62 patients with co-occurring current PTSD will be offered PE. Half of the 62 participants will be randomly assigned to a Prolonged Exposure with Contingency Management (PE+CM) condition that provides monetary-based incentives for attending the PE therapy sessions. The comparison condition will be assigned to a Prolonged Exposure (PE) condition without the attendance incentives intervention. The PE sessions will be scheduled once per week for 12 weeks, with a 12-week follow-up. Groups will be compared primarily on adherence to the PE schedule, improvement in PTSD symptoms, and rates of drug use (urine specimens, self-reported use). The study's three primary aims are to 1) Evaluate the efficacy of adding voucher-based attendance incentives to PE for PTSD to increase adherence in SUD patients in a methadone treatment program; 2) Evaluate the efficacy of adding voucher-based attendance incentives to PE for PTSD to reduce PTSD symptoms in SUD patients; and 3) Evaluate the effect of PE for PTSD on rates of drug use in SUD patients.

ELIGIBILITY:
Inclusion Criteria for Phase I (evaluation):

* positive screen for PTSD, as determined by score on the MPSS-R
* methadone maintenance for at least 4 weeks (to help ensure initial stabilization on methadone)
* at least 18 years of age

Inclusion criteria for Phase 2 (treatment):

* confirmation of current PTSD based on the Clinician-Administered PTSD Scale
* no psychiatric contraindications to PE (e.g., current suicidal/homicidal intent)
* clear memory for the traumatic event (e.g., flashbacks or re-experiencing the event)
* interest in receiving PE
* agree to sign release of information for any current psychiatric treatment providers outside of ATS
* agree to delay taking daily methadone dose on exposure therapy days until after session
* no history of prior exposure-based therapy for PTSD
* agree to audiotaping of therapy sessions

Exclusion Criteria:

* pregnancy
* acute medical problem that requires immediate and intense medical management (e.g., AIDS defining illness; active tuberculosis)
* presence of a formal thought disorder, delusions, hallucinations, or imminent risk of harm to self or others

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Prolonged Exposure session attendance | 12 weeks
  PE session attendance will be measured as the percent of participants completing a full course of PE and as a repeating dichotomous variable (weekly assessments of attended vs. unattended sessions).

SECONDARY OUTCOMES:
PTSD symptoms | 24 weeks
  Groups will be compared on PTSD symptoms (as measured by CAPS scores) collected at each assessment timepoint (baseline, week 6, week 12, week 24)
Drug use | 12 weeks
  Groups will be compared on weekly drug test results (presence/absence of drug) and on self-reported number of days using each drug during the 12-week treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Peirce, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services, Baltimore, Maryland, United States